CLINICAL TRIAL: NCT02146846
Title: Population Pharmacokinetics of Imatinib in CML Patients in Iran
Status: Terminated | Type: Observational
Sponsor: Kerman University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ehsan Mohajeri, Assistant of Pharmaceutics, Kerman University of Medical Sciences
Other Study IDs: Kerman-001-FOPPT
Record Dates: First submitted 2014-04-09; First posted 2014-05-26 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: cml
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Imatinib, CML: Patients with chronic myeloid leukemia who receive Imatinib as treatment in Iran entered in this study
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Patients with chronic myeloid leukemia who receive Imatinib as treatment
  Other Names: Glivec

SUMMARY:
The purpose of this study is to determine population Pharmacokinetics and differences and variation of pharmacokinetics parameters of Imatinib as a tyrosine kinase inhibitor in treatment of chronic myeloid leukemia patients in Iranian population.

DETAILED DESCRIPTION:
patients with chronic myeloid leukemia who receive Imatinib as treatment in Iran entered in this study then population pharmacokinetics parameters is determined.

ELIGIBILITY:
Inclusion Criteria:

* patient in chronic phase of myeloid leukemia
* no liver and renal failure

Exclusion Criteria:

* multiple dug treatment
* previous treatment of interferon
* patients in blast or accelerated phase

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with approved diagnosis of chronic myeloid leukemia taking Imatinib as treatment
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Percent of changes of AUC, trough Concentration from predicted values | Blood sampling are collected on atleast the 30th day of treatment at the following time: 1 hour before the dose and 1 hour after the dose
  The influence of patients' characteristic on the pharmacokinetics of Imatinib will be assessd.

CONTACTS AND LOCATIONS:
Overall Officials: ehsan mohajeri, Ph.D., Study Director — Department of pharmaceutics, Faculty of pharmacy, Kerman University of medical sciences
Locations (1):
- Shahid-Bahonar hospital, Kerman, Kerman, Iran